CLINICAL TRIAL: NCT05298371
Title: The Effect of Sitting and Standing Posture on Trunk Rotation in Patients With Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Burçin Akçay (Other)
Responsible Party: Sponsor-Investigator, Burçin Akçay, assistant professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Other Study IDs: B Akcay
Record Dates: First submitted 2022-03-06; First posted 2022-03-28 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Scoliosis Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with adolescent idiopathic scoliosis: Patients with AIS applying to Bandırma Onyedi Eylül University Physiotherapy and Rehabilitation Department will be included in this study.
  Individuals diagnosed with AIS, whose Cobb angle is between 20º -50º, who do not have any chronic disease requiring neurological or psychiatric medication, and who volunteered to participate in the study will be included. Individuals with any contraindications for exercise, previous spinal surgery, 6 or more curvature of the thoracic apex, mental problems, non-idiopathic scoliosis but with different causes will be excluded from the study.
  Interventions: Behavioral: Corrected Sitting postures; Behavioral: Natural / relaxed sitting postures; Behavioral: Corrected Standing posture; Behavioral: Natural / relaxed standing postures

INTERVENTIONS:
Behavioral: Corrected Sitting postures — Change after being in Corrected Sitting postures
Behavioral: Natural / relaxed sitting postures — Change after being in relaxed sitting postures
Behavioral: Corrected Standing posture — Change after being in Corrected Standing posture
Behavioral: Natural / relaxed standing postures — Change after being in relaxed standing postures

SUMMARY:
The aim of this study is to investigate the acute effect of activities of daily living on trunk rotation in patients with adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
Patients with AIS who applied to Bandırma Onyedi Eylül University Physiotherapy and Rehabilitation Department will be included in this study.

Individuals diagnosed with AIS, whose Cobb angle is between 20º -50º, who do not have any chronic diseases that require neurological or psychiatric medication, and who volunteer to participate in the study will be included. Individuals with any contraindications for exercise, previous spine surgery, thoracic apex curvature of 6 or more, mental problems, non-idiopathic scoliosis but with different causes will be excluded from the study.

To determine the demographic characteristics of the participants, age, gender, weight, height, presence of chronic disease, age at first diagnosis, exercise habits, treatments, and brace use will be questioned. The ATR will be used to measure degrees of trunk rotation to monitor the effects of treatment without radiographic evaluation.

On the first day, the demographic characteristics of the participants will be questioned, Cobb angles, Risser findings, and ATR degrees will be recorded. After the first day, all postural activities and measurements will be taken on different days (at least three days apart) not to affect the degrees of trunk rotation in patients with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with AIS between the ages of 10-35
* Cobb angle between 20º -50º,
* To be able to continue the program to be applied,
* Not having a chronic disease that requires the use of any neurological or psychiatric medication,
* The willingness of parents and/or patients to participate in the study.

Exclusion Criteria:

* The patient has any contraindications for exercise,
* Having had previous spine surgery,
* Having a curvature of 6 or more thoracic apex,
* Having any mental problems,
* The fact that scoliosis is not idiopathic but has arisen for different reasons (neurological, congenital, etc.)

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with adolescent idiopathic scoliosis.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Angle of trunk rotation (ATR) | Change from Baseline angle of trunk rotation at 5 minutes
  ATR can be used to monitor the effects of treatment without radiographic evaluation. ATR measurement is done using a special inclinometer called a scoliometer. The patient is asked to lean forward with the arms relaxed. The scoliometer is placed posteriorly and the degree observed at the point of greatest gimbosity is recorded.
Demographic Characteristics | Baseline
  Within the scope of the demographic information form, participants' age, gender, weight, height, presence of chronic diseases, age at which they were first diagnosed, exercise habits, treatments received, brace use will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Burçin Akçay, Study Director — Bandırma Onyedi Eylül University
Locations (1):
- Burçin Akçay, Balıkesir, Turkey (Türkiye)